CLINICAL TRIAL: NCT05607654
Title: The Mechanisms of Underlying Accelerated Repetitive Transcranial Magnetic Stimulation for Treatment-resistant Depression Via Reelin-Apoer2-NMDAR Pathway- Mediated Synaptic Plasticity
Brief Title: The Mechanisms of Underlying Accelerated Repetitive Transcranial Magnetic Stimulation for Treatment-resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 82271562
Record Dates: First submitted 2022-10-26; First posted 2022-11-07 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-09

CONDITIONS: Treatment-resistant Depression
Keywords: Treatment-resistant Depression; Repeated transcranial magnetic stimulation; Prefrontal-hippocampal circuit; Reelin; Synaptic plasticity
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active iTBS (Active Comparator): The active group of TRD will receive the accelerated intermittent TBS(iTBS).The iTBS cycles including 10 bursts of three pulses at 50 Hz were delivered in 2-second trains. Each iTBS session comprised 60 x 2 second trains, with an 8-second intertrain interval and total duration of 10-minutes.Treatment sessions were administered hourly 10 times a day totaling 18,000 pulses/day. Patients received this treatment protocol for 5 consecutive days (90,000 pulses in total).
  Interventions: Device: active iTBS
- sham rTMS (Sham Comparator): The sham group of TRD will receive sham rTMS stimulation.
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: active iTBS — Participants in the active stimulation group will receive the accelerated intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the neuronavigation system. Stimulation intensity will be standardized at 90% of RMT.
  Stimulation will be delivered to the L-DLPFC using an NTK-TMS-II100 TMS device,is compatible with the Brainsight TMS navigation system.
  Arms: active iTBS
Device: sham rTMS — The parameters in the sham arm will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: sham rTMS

SUMMARY:
In this project, the investigators evaluate an accelerated schedule of repetitive transcranial magnetic stimulation for treatment-resistant depression. The investigators focuse on participants' brain activity and blood markers (Reelin, Apoer2, NMDAR, BDNF, exosomes and so on) to deepen the understanding of the mechanism of accelerated rTMS for treatment-resistant depression.

DETAILED DESCRIPTION:
In this project, the investigator evaluate an accelerated schedule of repetitive transcranial magnetic stimulation for treatment-resistant depression. Patients were included in two groups and received an accelerated stimulation or sham treatment. The changes of neuroimaging and biomarkers at baseline, 5 days after treatment and 1 month after treatment are evaluated. The investigators focuse on participants' brain activity and blood markers (Reelin, Apoer2, NMDAR, BDNF, exosomes and so on) to deepen the understanding of the mechanism of accelerated rTMS for treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

1. The current episode met the DSM-5 diagnostic criteria for major depression in patients with first-episode or relapsed unmedicated depression without psychotic symptoms.
2. 24-item Hamilton Depression Scale (HAMD-24) ≥ 20.
3. Age 18-45 years, regardless of gender.
4. Right-handedness.
5. Han Chinese.
6. Signed a written informed consent, willing to participate in the study and be evaluated.

Exclusion Criteria:

1. Co-morbid other mental disorders, including: schizophrenia, mental retardation, substance dependence, etc.
2. Patients with metal objects in the body or with other contraindications to MRI scanning
3. Patients with severe or unstable somatic diseases
4. Women during pregnancy or lactation, and women of childbearing age with positive urine HCG test results during the screening period
5. Other conditions that, in the opinion of the investigator, exist that make participation in this clinical trial inappropriate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in remission rate of Hamilton Depression Scale (24-items) (HAM-D24) score after treatment. | Baseline, 5-day, 1-month
  The Hamilton Depression Scale (24-items) (HAM-D24), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4.
  Remission is defined as HAM-D24 ≤8.

SECONDARY OUTCOMES:
Change in response rate of Hamilton Depression Scale (24-items) (HAM-D24) score after treatment. | Baseline, 5-day, 1-month
  The Hamilton Depression Scale (24-items) (HAM-D24), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4.
  Response is defined as a reduction of >/=50% of HAM-D24 baseline score.
Change in the rate of Beck Scale of Suicidal Ideation score after treatment. | Baseline, 5-day, 1-month
  Beck Scale of Suicidal Ideation(BSI) is a 21-item self-report instrument that detects and measures the intensity of a patient's specific attitudes, behaviors, and suicide plans during the past week.
Change in the rate of Hamilton Anxiety Scale score after treatment. | Baseline, 5-day, 1-month
  Hamilton Anxiety Scale (HAMA) is a 17 item diagnostic questionnaire used to measure the severity of anxiety episodes in patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No